CLINICAL TRIAL: NCT03655158
Title: The Effects of Ozone Therapy on Wound Healing After Gingivectomy Operations: a Controlled Clinical Study
Brief Title: The Effects of Ozone Therapy on Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zekeriya Tasdemir, Principal investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Zektaşdemir
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Wound Heal

STUDY DESIGN:
Intervention Model Description: Split- mouth placebo controlled design (right quadrants of the surgical areas were assigned to receive ozone therapy in all patients. As placebo application, left quadrants received regular air from the ozone generator)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: placebo applications were performed to mask participant
  investigator who applied ozone, did not evaluate the healing
  Investigator who evaluate the healing, did not know the control and test sides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone group (Experimental): After gingivectomy and gingivoplasty, right quadrants of the surgical areas were assigned to receive ozone therapy in all patients
  Interventions: Device: ozone device ( Ozonytron XL )
- non-ozone group (No Intervention): placebo application, left quadrants received regular air from the ozone generator.

INTERVENTIONS:
Device: ozone device ( Ozonytron XL ) — The adjustment of the ozone generator was %75 power for 30 seconds (75 ug/ml) based on manufacturer's instructions
  Arms: ozone group

SUMMARY:
the aim of present study was to evaluate effects of ozone therapy on wound healing after gingivectomy and gingivoplasty operations as a model of secondary wound healing.. Twenty three systemically healthy individuals participated in this study. Ozone was applied immediately after surgery, at 1st day and 3rd day after gingivectomy surgery. In the photographs of the wounds, the difference in color were evaluated and measurements were performed at the baseline, 3rd, 7th, 14th days after surgery.

DETAILED DESCRIPTION:
Although ozone therapy has often been tried in medical science and has become more popular due to its antimicrobial, biocompatibility and healing properties, the effects of ozone therapy on surgeries that heals with secondary intention were not studied. In the lights of these informations, the aim of present study was to evaluate effects of ozone therapy on wound healing after gingivectomy and gingivoplasty operations as a model of secondary wound healing. Twenty three systemically healthy individuals participated in this study. All periodontal examinations were performed by one experienced examiner and non-surgical periodontal treatment of the patients were performed within two weeks after initial examination by the same clinician.Gingivectomy and gingivoplasty operations were performed by another examiner who was unaware of the study protocol.After gingivectomy and gingivoplasty, right quadrants of the surgical areas were assigned to receive ozone therapy in all patients. Ozone therapy was also performed by an experienced periodontist. As placebo application, left quadrants received regular air from the ozone generator.Postoperative pain was assessed at 3rd, 7th, 14th days after surgery with a visual analog scale At baseline and 3rd, 7th, 14th days after surgery, surgical area was disclosed by a plaque disclosing solution to visualize the epithelization degree of the surgical areas. Solution provided a clear vision to distinguish normal gingiva from the areas in which the gingival epithelium is absent, abraded or lacking sufficient keratinization. In order to evaluate epithelization degree of the wounds, standardized photographs were taken from each patient.In the photographs of the wounds, the difference in color were evaluated and darkly stained areas were considered as lack of enough epithelization. These measurements were performed at the baseline, 3rd, 7th, 14th days after surgery. The determinations were done by a calibrated examiner who was blind to test and control sites

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years of age
* systemically healthy
* non-smokers
* no medications taken for 6 months
* no pregnancy and lactation
* no contraindications for periodontal surgery
* no gingivectomy or mucogingival surgical history in the lower incisor region.

Exclusion Criteria:

* <18 and > 35 years of age
* systemical disease
* smoking and alcohol consumption
* medications taken for 6 months
* pregnancy and lactation
* contraindications for periodontal surgery
* gingivectomy or mucogingival surgical history in the lower incisor region.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
wound healing change | At baseline and 3rd, 7th, 14th days after surgery, wound healing evaluation were performed.
  surgical area was disclosed by a plaque disclosing solution to visualize the epithelization degree of the surgical areas. Solution provided a clear vision to distinguish normal gingiva from the areas in which the gingival epithelium is absent, abraded or lacking sufficient keratinization. In order to evaluate epithelization degree of the wounds, standardized photographs were taken from each patient

SECONDARY OUTCOMES:
Pain change | Postoperative pain was assessed at 3rd, 7th, 14th days after surgery
  Visual analog scale was used for the pain assesment. On the scale, the left end of the graphic represented the absence of pain (score 0) and the right end represented the most severe pain (score 10).

CONTACTS AND LOCATIONS:
Overall Officials: Zekeriya Taşdemir, Phd, Principal Investigator — TC Erciyes University
Locations (1):
- Zekeriya Taşdemir, Kayseri, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided